CLINICAL TRIAL: NCT02475551
Title: A Phase II Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of Intravenous Ascending Doses of IdeS in Kidney Transplantation
Brief Title: Study to Evaluate the Safety, Tolerability, Efficacy and PK of IdeS in Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Collaborators: Uppsala University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-HMedIdeS-03
Record Dates: First submitted 2015-06-05; First posted 2015-06-18 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): IdeS as a single infusion
  Interventions: Drug: IdeS

INTERVENTIONS:
Drug: IdeS — Intravenous infusion

SUMMARY:
This study will assess the safety and efficacy of IdeS in the transplantation setting. Each patient will receive one dose of IdeS. If the crossmatch test is negative at the time of transplantation, the patient will be transplanted with a kidney from a deceased or living donor. The starting dose will be 0.25 mg/kg BW, given as a single intravenous infusion prior to surgery.

DETAILED DESCRIPTION:
This study will assess the safety and efficacy of the IgG degrading cysteine protease IdeS in the transplantation setting. Patients with DSAs will be treated with IdeS prior to transplantation. Each patient will receive one dose of IdeS. If the crossmatch test is negative after IdeS treatment, the patient will be transplanted with a kidney from a deceased or living donor. Two to four dose groups are planned. Each group will contain 2 patients with the possibility to extend the group to up to 4 patients per group if required for safety and/or efficacy evaluation. The starting dose will be 0.25 mg/kg BW, given as a single intravenous infusion prior to surgery with the possibility to increase the dose in higher dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CKD and in dialysis with preformed anti-HLA antibodies (non-DSA, DSA or both), negative T-CDC CXM and at least one antibody MFI > 3000

Exclusion Criteria:

* Prior malignancy within 2 years excluding adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ and prostate cancer Gleason <6 and prostate-specific antigen (PSA) <10 ng/mL.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV
* Clinical signs of ongoing infectious disease.
* Severe other conditions requiring treatment and close monitoring, e.g. cardiac failure > New York Heart Association (NYHA) grade 3, unstable coronary disease or oxygen dependent chronic obstructive pulmonary disease (COPD)
* History of any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at increased risk because of participation in the study, or influence the results or the patient's ability to participate in the study
* Hypogammaglobulinemia defined as any values of P-total IgG less than 3 g/L
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to IdeS (e. g streptokinase and/or staphylokinase)
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 4 months of the first administration of investigational product in this study.
* Patients consented and screened but not dosed in previous studies are not excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
safety | 6 months
  Adverse events, clinical laboratory tests, vital signs and ECGs

SECONDARY OUTCOMES:
Efficacy (mean fluorescent intensity (MFI) of less than 1100 as measured in an single antigen bead (SAB) assay) | 24 hours
  Efficacy defined as the IdeS dosing scheme resulting in anti human leucocyte antigen (HLA) antibody levels which are acceptable for transplantation, measured as an mean fluorescent intensity (MFI) of less than 1100 as measured in an single antigen bead (SAB) assay, within 24 hours from dosing

CONTACTS AND LOCATIONS:
Overall Officials: Lena Winstedt, PhD, Study Director — Hansa Biopharma AB
Locations (1):
- Hansa Medical AB, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernando SC, Polkinghorne KR, Lim WH, Mulley WR. Early Versus Late Acute AMR in Kidney Transplant Recipients-A Comparison of Treatment Approaches and Outcomes From the ANZDATA Registry. Transplantation. 2023 Nov 1;107(11):2424-2432. doi: 10.1097/TP.0000000000004700. Epub 2023 Jun 16. PMID 37322595
- [Derived] Jordan SC, Lorant T, Choi J, Kjellman C, Winstedt L, Bengtsson M, Zhang X, Eich T, Toyoda M, Eriksson BM, Ge S, Peng A, Jarnum S, Wood KJ, Lundgren T, Wennberg L, Backman L, Larsson E, Villicana R, Kahwaji J, Louie S, Kang A, Haas M, Nast C, Vo A, Tufveson G. IgG Endopeptidase in Highly Sensitized Patients Undergoing Transplantation. N Engl J Med. 2017 Aug 3;377(5):442-453. doi: 10.1056/NEJMoa1612567. PMID 28767349